CLINICAL TRIAL: NCT05359289
Title: Effects of Forest Therapy on Cognitive Performance and Mental Health in Older Adults
Brief Title: Effects of Forest Therapy on Cognitive Performance and Mental Health in Older Adults Health in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); National Taiwan University (Other); National Taiwan Science Education Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202105HM079
Record Dates: First submitted 2022-04-07; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-08

CONDITIONS: Forest Therapy for Cognition
Keywords: forest therapy; successful ageing; physical and mental health; cognitive health; senior fitness; clinic trial; brain imaging
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Forest therapy training (Experimental): Participants will expect to have an improvement of cognitive functions via a serial nature-based therapy/intervention.
  Interventions: Behavioral: Forest therapy training
- Senior fitness training (Active Comparator): Participants will expect to have an improvement of cognitive functions through a structural senior fitness program.
  Interventions: Behavioral: Senior fitness training
- Board Games (Placebo Comparator): Participants will play boards games under a schedule matching the Experimental and Active Comparator arms.
  Interventions: Behavioral: Board Games

INTERVENTIONS:
Behavioral: Forest therapy training — Participants will experience nature-based interventions including forest hiking, horticultural therapy and green wellness activities for their mental health and physical conditions.
  Arms: Forest therapy training
Behavioral: Senior fitness training — The fitness program includes physics fitness of stamina, coordination and aerobic exercise in 12 weeks. Participants will join the senior fitness program including physical fitness, aerobic exercise and exercise prescription during the 12 weeks program.
  Arms: Senior fitness training
Behavioral: Board Games — Participants will play board games with each other.
  Arms: Board Games

SUMMARY:
In Taiwan, aging is happening at a fast pace. The Taiwan Ministry of Interior officially announced that Taiwan will become an aged society in April 2018 and is expected to transition into a hyper-aged society within eight years. Critically, scholars recognize that optimizing cognitive activity and wellbeing influences quality of life in a late life which in turn is a key factor for successful aging. To alleviate the social and economic impact of aging, as well as impact on families, there is a need for studying anti-aging approaches. The World Health Organization suggests that the general public should have a healthy lifestyle which includes participating in activities for physical health, as well as cognitive and mental health involving maintaining social interactions. This present research is part of a broader integrated program in which the purpose is to promote and study the efficacy of forest therapy on physical health, and cognitive and mental health in older adults. The study site is located at the National Taiwan Science Education Center (NTSEC) which includes wetlands, waterfronts, green-spaces and urban parks. The investigators will evaluate two types of interventions for participants, "forest therapy program" and "fitness program" for older adults. The study approach applies a between-subjects and pretest-posttest design. The investigators will collect participants' physical data, psychological responses, and cognitive performance in the course of both programs. By comparing these data before and after the intervention programs, the investigators seek to understand the both programs' effects on physical health, and cognitive and mental health.

DETAILED DESCRIPTION:
In Taiwan, aging is happening at a fast pace. The Taiwan Ministry of Interior officially announced that Taiwan will become an aged society in April 2018 and is expected to transition into a hyper-aged society within eight years. Critically, scholars recognize that optimizing cognitive activity and wellbeing influences quality of life in a late life which in turn is a key factor for successful aging. To alleviate the social and economic impact of aging, as well as impact on families, there is a need for studying anti-aging approaches. The World Health Organization suggests that the general public should have a healthy lifestyle which includes participating in activities for physical health, as well as cognitive and mental health involving maintaining social interactions. This present research is part of a broader integrated program in which the purpose is to promote and study the efficacy of forest therapy on physical health, and cognitive and mental health in older adults. The study site is located at the National Taiwan Science Education Center (NTSEC) which includes wetlands, waterfronts, green-spaces and urban parks. The investigators will evaluate two types of interventions for participants, "forest therapy program" and "fitness program" for older adults. The study approach applies a between-subjects and pretest-posttest design. The investigators will collect participants' physical data, psychological responses, and cognitive performance in the course of both programs. By comparing these data before and after the intervention programs, the investigators seek to understand the both programs' effects on physical health, and cognitive and mental health. In addition, the investigators will elucidate the efficacy of the forest therapy program through measurement of the changes in physical, cognitive, and mental health performance and status indicators. The forest therapy and fitness programs at National Taiwan Science Education Center (NTSEC), along with a robot programming training and tinkering activities that are part of the broader project, acts as a public education and service window towards addressing cognitive aging issues in Taiwan. It should be further noted that this will be a critical platform for obtaining ecological research data on a novel class of cognitive interventions for cognitive aging using psychological and brain imaging techniques to bridge critical neural mechanistic knowledge gaps.

ELIGIBILITY:
Inclusion Criteria:

* Literate in Mandarin and Taiwanese.
* Willing to participate entirely in this research.
* Age > 65.

Exclusion Criteria:

* Participated in cognitive-related training in the past two months.
* Diagnosed with mild cognitive impairment(MCI)
* Severe psychological or behavioral disorder that would seriously interfere with the progress of activity.
* Severe hearing Impairments or visual Impairment
* History of degenerative cognitive disorders, Organic Mental Disorders, Brain Dysfunction, Psychogenic neurosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Changes of neural functional activity during inferential processing | week 0, week 12
  Participants will undergo a Rule Inference fMRI task to infer underlying rules that map color configurations of circles in a triangular arrangement to a target color category within as few tries as possible under active or passive conditions.The goal for participants will be to infer the cue-category association rules using as few cues as possible. The primary outcome measure here is the degree of neural response estimate change in blood oxygen level dependent (BOLD)signal pre- and post-intervention.
Changes of overall accuracy during inferential processing | week 0, week 12
  Changes from pre- to post-intervention in participant overall accuracy in identifying latent rules in the Rule Inference fMRI task.
Changes of learning rate during inferential processing | week 0, week 12
  Changes from pre- to post-intervention in participant number of trials to criterion in the Rule Inference fMRI task.
Changes of strategic performance during inferential processing | week 0, week 12
  Changes from pre- to post-intervention in participant coefficients of expression of modeled response strategies in the Rule Inference fMRI task will be assessed.
Changes in the Montreal Cognitive Assessment (MoCA) score | week 0, week 12
  Pre- to post-intervention changes in participant MoCA score. Score range from 0 to 30 with higher scores indicating better cognitive ability.
Change in Wechsler Memory Scale III Logical Memory I & II | week 0, week 12
  Score range 0 - 75. Higher score indicates better verbal episodic memory.
Change in Wechsler Memory Scale III Face Memory | week 0, week 12
  Score range 0 - 48. Higher score indicates better visual face memory.
Change in Wechsler Memory Scale III Verbal Paired Memory | week 0, week 12
  Score range 0 - 32. Higher score indicates better verbal memory and learning.
Change in Wechsler Memory Scale III Family Pictures I & II | week 0, week 12
  Score range 0 - 64. Higher score indicates better visual memory and learning.
Change in Wechsler Memory Scale III Word Lists I & II | week 0, week 12
  Score range 0 - 36. Higher score indicates better verbal memory and learning. For II, recall score range is 0 to 8; recognition score range is 0 to 24.
Change in Wechsler Memory Scale III Visual Reproduction I & II | week 0, week 12
  Score range 0 - 104. Higher score indicates better visual memory. For II, recall score range is 0-104; recognition score range is 0-48.
Change in Wechsler Memory Scale III Spatial Span | week 0, week 12
  Score range 0 - 32. Higher score indicates better spatial memory. range is 0-48.
Change in Wechsler Memory Scale III Digit Span | week 0, week 12
  Score range 0 - 32. Higher score indicates better auditory memory.
Change in Wechsler Adult Intelligence Scale III Vocabulary | week 0, week 12
  Score range 0 - 66. Higher score indicates better vocabulary.
Change in Wechsler Adult Intelligence Scale III Digit Symbol | week 0, week 12
  Score range 0 - 133. Higher score indicates better processing speed.
Change in Wechsler Adult Intelligence Scale III Block Design | week 0, week 12
  Score range 0 - 68. Higher score indicates better visual processing.
Change in Wechsler Adult Intelligence Scale III Arithmetic | week 0, week 12
  Score range 0 - 22. Higher score indicates better mathematical computation ability.
Change in Wechsler Adult Intelligence Scale III Matrix Reasoning | week 0, week 12
  Score range 0 - 26. Higher score indicates better reasoning.
Change in the Profile of Mood States(POMS) | week 0, week 12
  Pre- to post-intervention changes in participant POMS score. Score range from 0 to 24 with higher scores indicating the level of each mood States, as tension-anxiety, anger-hostility, depression-dejection, fatigue-inertia, confusion-bewilderment, vigor-activity.
Change in State-Trait Anxiety Inventory(STAI) | week 0, week 12
  Pre- to post-intervention changes in participant STAI score. Score range from 0 to 80 with higher scores indicating higher anxiety level.
Change in Chinese Word Remote Associate Task(CWRAT) | week 0, week 12
  Pre- to post-intervention changes in participant CWRAT score. Score range from 0 to 80 with higher scores indicating better creativity.
Change in Diastolic Blood Pressure(DBP) and Systolic Blood Pressure(SBP) | week 0, week 12
  Pre- to post-intervention changes in participant blood pressure. Normal SBP of an adult under 120 mmHg and normal DBP under 80 mmHg with lower pressure indicating better health.
Change in heart rate | week 0, week 12
  Pre- to post-intervention changes in participant heart rate. The normal heart rate of an adult beats between 60 to 100 times per minute, with lower times indicating better health.
Change in heart rate variability (HRV) | week 0, week 12
  Changes from pre- to post-intervention in participant HRV. In sympathetic nervous system, with lower ratio of Low/High Frequency and higher high Frequency indicating better relaxation.
Change in Body Mass Index(BMI) | week 0, week 12
  Changes from pre- to post-intervention in participant Body Mass Index.
Change in Waist-Hip Ratio | week 0, week 12
  Changes from pre- to post-intervention in participant Waist-Hip Ratio.
Change in 30s arm curl test | week 0, week 12
  Changes from pre- to post-intervention in participant 30s arm curl test, with higher times indicating better strength.
Change in 30s chair stand test | week 0, week 12
  Changes from pre- to post-intervention in participant 30s chair stand test, with higher times indicating better endurance.
Change in back scratch test | week 0, week 12
  Changes from pre- to post-intervention in participant 30s back scratch test, with higher times indicating better upper limb flexibility.
Change in chair sit-and-reach test | week 0, week 12
  Changes from pre- to post-intervention in participant 30s chair sit-and-reach test, with higher times indicating better lower limb flexibility.
Change in Seated Up- and- Go Test | week 0, week 12
  Changes from pre- to post-intervention in participant Seated Up- and- Go Test, with fewer time indicating better dynamic balance and agility.
Change in 2-minute step test | week 0, week 12
  Changes from pre- to post-intervention in participant Seated Up- and- Go Test, with higher times indicating better cardiorespiratory fitness.

SECONDARY OUTCOMES:
Changes of neural functional activity during resting-state | week 0, week 12
  Brain functional activity measured using fMRI during rest with eyes-open

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Pin Yu, Ph.D., Principal Investigator — National Taiwan University
Locations (2):
- Taiwan (2):
  - School of Forestry and Resource Conservation, National Taiwan University, Taipei
  - National Taiwan Science Education Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared include anonymized neuropsychological assessment scores, cognitive behavioral performance scores, brain imaging data that have been published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available 1 year after primary results are published by the central research team. Data are anticipated to be available for sharing for an indefinite period after the above criteria is met.
Access Criteria: Data sharing will be done based direct requests and on case-by-case evaluation for appropriateness. Use of shared data will require agreement on appropriate citation of data sources at least or authorship inclusion or acknowledgement.